CLINICAL TRIAL: NCT01290185
Title: Improving the Success Rate of Continuous Peripheral Nerve Blocks Using a Novel Coiled Catheter
Brief Title: Coiled Catheters for Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Cedric Luyet, MD, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Luyet Coiled Catheters
Record Dates: First submitted 2011-01-31; First posted 2011-02-04 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Arthritis
Keywords: Arthroplasty; Pharmacol Nerve Block
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coiled Catheter (Experimental): Placement of the coiled catheter for continuous infusion of local anesthetics close to the femoral nerve: To place coiled catheters ab 18-gauge Tuohy needle (Sonoline Curl Catheter Set, Pajunk® Medizintechnologie GmbH, Geisingen, Germany) of 8 cm length is placed adjacent to the nerve by ultrasound guidance and nerve stimulator control. At this position and after injection of 5 ml dextrose 5% in water to dilate the space the coiled catheter is blindly advanced 2 cm through the needle and the final position verified with ultrasound.
  Interventions: Device: Placement of different catheters for continuous nerve block
- Conventional stimulating Catheter (Active Comparator): For the control group a conventional stimulating catheter is placed adjacent to the femoral nerve as follows: To place the simulating catheter an 18-gauge Tuhoy needle s placed adjacenit to the nerve by ultrasound guidance. At this position a stimulation catheter is introduced through the needle and stimulated with a decreasing current from 1 mA to 0.4 mA, with a pulse width 0.1ms to verify the appropriate motor response of the quadriceps muscle. The catheter is slowly advanced 3 cm beyond the needle tip under continuous electric stimulation using a current that is subsequently adapted according to the motor response achieved. If muscles twitches disappear during catheter placement at a current above 1 mA, either the catheter or the needle are manipulated until muscle twitches reappear.
  Interventions: Device: Placement of different catheters for continuous nerve block

INTERVENTIONS:
Device: Placement of different catheters for continuous nerve block — Placement different catheters adjacent to the femoral
  Other Names: Sonoline Curl Catheter Set, Pajunk; StimuCath; Arrow International

SUMMARY:
Major orthopaedic surgery is painful and requires safe and effective postoperative analgesic therapy. The successful use of continuous peripheral nerve blocks provides sustained analgesia while minimizing the need for opioid analgesics throughout the postoperative period and avoiding the side effects associated with central neuraxial techniques. Excellent analgesia can be maintained and opioid-related side effects avoided allowing improved rehabilitation. However using existing methods a failure rate of >20% significantly limits the analgesic benefits in a substantial proportion leading to uncontrolled pain and side effects of opioid analgesics.

A major concern with the use of continuous peripheral nerve blocks is difficulty in placement of the catheters close enough to the nerve to allow for effective local anaesthetic spread and therefore analgesia. The benefit of ultrasound to precisely place needles adjacent to nerves and increase efficacy of block success is undisputed. However ultrasound is of less help in accurately placing catheters. Indeed the final position of the catheter tip is not predictable and can be inadequate in 10%-50% of cases. The explanation for that is the material in currently used catheters is stiff and designed to avoid kinking. Unfortunately this same stiffness often leads to inadequate placement of the catheter tip. We have developed a catheter which coils up as soon as it is advanced beyond the needle tip, thus allowing the catheter tip to remain close to the initial needle tip position and therefore the nerve. The aim of this prospective randomized double blind controlled study is to determine the effectiveness of this new catheter in comparison with standard of care methods for continuous femoral nerve block commonly used after total knee arthroplasty. The primary outcome measure will be the incidence of catheter related block failure 24 hours after surgery. Our hypothesis is that the coiled catheter will significantly improve the efficacy of continuous femoral nerve block as compared to existing techniques.

DETAILED DESCRIPTION:
Aims of the study The aim is to determine the effectiveness of a the coiled catheter for continuous peripheral nerve block after total knee arthroplasty based on secondary block failures compared to the secondary block failures of the conventional, currently used stimulating catheters.

Study design The trial is a prospective single-centre randomized double-blinded controlled trial. Patients will be randomized to (1) use of conventional stimulating catheters or (2) to use of a coiled catheter.

Patient population Adult patients of at least 18 years of age undergoing unilateral knee arthroplasty, under spinal anaesthesia will be recruited in this randomized double blind controlled trial.

Inclusion criteria: Ability to provide informed consent, understanding of the possible local anaesthetic-related complications, and understanding of the study protocol.

Exclusion criteria: Any contraindication to peripheral nerve block, allergy to local anaesthetics, infection near the insertion site, ASA classification IV or V, pregnancy, chronic opioid analgesic therapy (>30mg morphine equivalent per day), coagulopathy, known hepatic or renal insufficiency, peripheral neuropathy and patient refusal.

ELIGIBILITY:
Inclusion Criteria:

Ability to provide informed consent, understanding of the possible local anaesthetic-related complications, and understanding of the study protocol.

Exclusion Criteria:

Any contraindication to peripheral nerve block, allergy to local anaesthetics, infection near the insertion site, ASA classification IV or V, pregnancy, chronic opioid analgesic therapy (>30mg morphine equivalent per day), coagulopathy, known hepatic or renal insufficiency, peripheral neuropathy and patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Secondary block failure rate | 24 hours after intervention (i.e. catheter placement)
  The primary outcome measure will be the presence or absence of analgesia (loss of temperature sensation in the femoral nerve distribution) on postoperative day 1 at 24 hours after placement of the catheter.
  Secondary block failure rates are defined as presence of temperature sensation in the sensory distribution of the femoral nerve i.e.: anterior aspect of the thigh and anteromedial lower leg.

SECONDARY OUTCOMES:
Catheter placement | 1 Minute after Catheter placement
  1. Technical difficulty of catheter placement: a. Number of attempts to place the catheter. b. lowest nerve stimulator output current at the final position of the catheter.
  2. Total time taken to place the catheter.
  3. Primary block failures as evaluated during the first 20 minutes after injection of Mepivacaine 1% through the catheters; defined as only partial or absent sensory or motor block in the sensory distribution of the femoral nerve as is: anterior aspect of the thigh and strength of quadriceps muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Colin J McCartney, M.D., Study Director — Sunnybrook Health Sciences Centres, Toronto; Cédric Luyet, M.D., Principal Investigator — Sunnybrook Health Sciences Centres, Toronto
Locations (1):
- Sunnybrook Health Sciences Centres, Holland Orthopedic and Arthritic Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Luyet C, Seiler R, Herrmann G, Hatch GM, Ross S, Eichenberger U. Newly designed, self-coiling catheters for regional anesthesia--an imaging study. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):171-6. doi: 10.1097/AAP.0b013e31820d431a. PMID 21270719